CLINICAL TRIAL: NCT00748605
Title: A Double-Blind, Multi-Center, Randomized, Parallel-Group, Yearlong Study to Assess the Efficacy and Safety of 0 or 1600 mg/Day of S-2367 Administered Orally Once Daily With an Initial 6-Week Low Calorie Diet in Obese Males and Females
Brief Title: Phase IIb One Year Efficacy and Safety Study of S-2367 in Obese Subjects With Initial 6-Week Low Calorie Diet
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0702A2824 revised
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity | interventions — Caloric Restriction; Apoptosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): S-2367 placebo + LCD (Low Calorie Diet) +RCD (Reduced Calorie Diet)
  Interventions: Drug: S-2367 Placebo; Other: LCD (low calorie diet); Other: RCD (reduced calorie diet)
- S-2367 1600 mg q.d. 54 weeks (Experimental): S-2367 placebo + LCD for 6 weeks and 1600 mg S-2367 + RCD for 54 weeks
  Interventions: Drug: S-2367 Placebo; Drug: S-2367 1600 mg q.d. 54 Weeks; Other: LCD (low calorie diet); Other: RCD (reduced calorie diet)
- S-2367 1600 mg q.d. 60 weeks (Experimental): S-23671600 mg q.d. + LCD for 6 weeks and S-2367 1600 mg q.d + RCD for 54 weeks
  Interventions: Drug: S-2367 1600 mg q.d. 60 weeks; Other: LCD (low calorie diet); Other: RCD (reduced calorie diet)

INTERVENTIONS:
Drug: S-2367 Placebo — Four placebo tablets (total dose = 0 mg/day S-2367) administered orally once daily with AM (ante meridiem) meal while on both LCD (low calorie diet for 6 weeks) and RCD (reduced calorie diet for 54 weeks) for a total of 60 weeks
  Arms: Placebo; S-2367 1600 mg q.d. 54 weeks
Drug: S-2367 1600 mg q.d. 54 Weeks — Four 400 mg S- 2367 tablets (total dose = 1600 mg/day S-2367) administered orally once daily with AM meal while on RCD for a total of 54 weeks
  Other Names: Velneperit
  Arms: S-2367 1600 mg q.d. 54 weeks
Drug: S-2367 1600 mg q.d. 60 weeks — Four 400 mg S- 2367 tablets (total dose = 1600 mg/day S-2367) administered orally once daily with AM meal while on both LCD and RCD for a total of 60 weeks
  Other Names: Velneperit
  Arms: S-2367 1600 mg q.d. 60 weeks
Other: LCD (low calorie diet) — A low calorie diet was utilized during the first 6 weeks of the study
Other: RCD (reduced calorie diet) — A reduced calorie diet was used during the last 54 weeks for the study

SUMMARY:
1. To evaluate the weight loss effect of 1600 mg/day S-2367 administered orally once daily with the morning meal after a 6-week low calorie diet (LCD) of 950 kcal/day with or without S-2367 followed by 54 weeks while on a 800 kcal deficit reduced calorie diet (RCD) compared with placebo in medically stable and otherwise healthy obese male and female subjects
2. To evaluate the safety and tolerability of 1600 mg/day S-2367 administered orally once daily with the morning meal after a 6-week LCD with or without S-2367 followed by 54 weeks on a RCD compared with placebo in medically stable and otherwise healthy obese male and female subjects
3. To evaluate the steady-state/trough pharmacokinetics of 1600 mg/day S-2367 administered orally once daily with the morning meal after a 6-week LCD with or without S-2367 followed by 54 weeks on a RCD in obese male and female subjects
4. To evaluate the weight loss effect of 1600 mg/day S-2367 administered orally once daily with the morning meal during an initial 6-week LCD compared with placebo in medically stable and otherwise healthy obese male and female subjects

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 65 years of age and body mass index between 30.0 to 45.0 kg/m2, inclusive, and a weight that has not fluctuated by more than 3% for the last 3 months
* Medically stable for 3 months prior to Visit 1 and in otherwise good health, with no clinically significant findings from medical history, physical examination, 12-lead electrocardiograms (ECGs), and vital signs
* Clinical laboratory evaluations (including clinical chemistry [fasted at least 8 hours], complete blood count, urinalysis, including creatine phosphokinase, amylase, lipase, lipid profile, insulin, Homeostatic Model Assessment of Insulin Sensitivity Index, hemoglobin A1c, thyroid stimulating hormone, free thyroxine, cortisol, iron, and ferritin) within the reference range for the test laboratory, unless deemed not clinically significant by the investigator
* Males will be sterile or agree to use an approved method of contraception. Some of the approved methods of contraception for males includes a surgically sterile (for at least 3 months prior to Visit 1) female sexual partner; a postmenopausal (for at least 1 year since last menstrual cycle) female sexual partner; a female sexual partner who uses (for at least previous 3 months prior to Visit 1 and during study) oral, implantable, transdermal, or injectable oral contraceptives; or use of the following double-barrier method: male condom with spermicide
* Females will be non-pregnant, non-lactating, and either postmenopausal for at least 1 year since last menstrual period, surgically sterile for at least 3 months prior to Visit 1, or agree to use an approved method of contraception. Some of the approved methods of contraception for females include a sterile (for at least 3 months prior to Visit 1) male sexual partner; use of oral, implantable, transdermal, or injectable oral contraceptives; or use of one of the following double-barrier methods: intrauterine device with spermicide, diaphragm with spermicide, cervical cap with spermicide, female condom with spermicide, or a male condom with spermicide by the male sexual partner
* Able to understand and willing to sign an informed consent form and comply with all study procedures

Exclusion Criteria:

* History or clinical manifestations of significant metabolic, hepatic, immunological (e.g., human immunodeficiency virus/ acquired immunodeficiency syndrome), renal, hematological, pulmonary, cardiovascular, gastrointestinal (GI), urological, neurological, or psychiatric disorders
* History or presence of an abnormal ECG, which in the investigator's opinion, is clinically significant
* History or evidence of a psychological disorder, other than stable or controlled anxiety or depression, including but not limited to the schizophrenias. Treatment with an antidepressant or anxiolytic drug(s) will be permitted if the dose and form has remained stable for at least the previous 3 months and the medication is not precluded/ excluded by this protocol because of potential effects on body weight and is not expected to change during the remainder of this clinical protocol
* History or evidence of an eating disorder with a compensatory behavior such as "purging bulimia nervosa" or "non-purging bulimia nervosa"
* History of obesity of endocrine origin
* History of Type 1 or Type 2 diabetes mellitus
* Clinically significant hypertension defined as blood pressure > 160/90 mm Hg for either the systolic or diastolic values in either the untreated or treated state
* Clinically significant GI history or surgery. NOTE: Appendectomy and cholecystectomy will be allowed
* Gastric bypass surgery, stomach banding surgery, or any other surgical procedure(s) that attempt to promote/aid weight loss
* History of polycystic ovarian syndrome
* History of fenfluramine or dexfenfluramine or "fen-phen" administration with abnormal findings on echocardiograms at the time of "fen-phen" discontinuation
* History of participation in any weight loss program within 3 months prior to Visit 1
* History of body weight loss or gain greater than 3% within 3 months prior to Visit 1
* History of alcoholism or drug addiction/ substance abuse within 1 year prior to Visit 1
* History of any tobacco-containing or nicotine-containing product use within 1 year prior to Visit 1
* Participation in any other investigational study drug trial in which receipt of investigational study drug occurred within 3 months prior to Visit 1
* Previous use or participation in a study of S-2367 or any other neuropeptide Y5 agonist or antagonist
* Participation in any weight loss medication/product study in which receipt of weight loss medication/product occurred within 3 months prior to Visit 1
* Use of any prescription or non-prescription over-the-counter (OTC) medication/product or herbal/phytotherapeutic/plant-derived medications/products within 3 months prior to Visit 1 that is intended to induce weight loss, appetite suppression, weight control, or treat obesity
* Use of chronic medications/products within 3 months prior to Visit 1 or during the study that are known to cause weight gain. The list includes but is not limited to amitriptyline (Elavil), paroxetine (Paxil), setraline (Zoloft), and mirtazepine (Remeron)
* Use of any prescription or non-prescription OTC medications/products within 1 month prior to Visit 1, unless deemed acceptable by the investigator.
* Donation of blood or blood products 3 months prior to Visit 1 or during the entire study
* Any acute or chronic condition that, in the opinion of the investigator, would limit the subject's ability to complete and/ or participate in this clinical study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 842 (Actual)
Dates: Start 2007-06; Primary Completion 2008-11 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
The change in body weight over the 60-week active therapy phase of the study | 60 weeks

SECONDARY OUTCOMES:
Change in body composition: calculated body mass index, waist circumference, hip circumference, and calculated waist-to-hip ratio | Throughout the study
Steady-state/trough pharmacokinetic analysis | After 9, 18, 30, 42, and 60 weeks of study drug treatment
Safety and tolerability of S-2367: treatment emergent adverse events, clinical laboratory data, vital signs, and 12-lead electrocardiogram parameters at each visit | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (40):
- United States (40):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Phoenix, Arizona
  - Fountain Valley, California
  - San Diego, California
  - San Francisco, California
  - Waterbury, Connecticut
  - Jacksonville, Florida
  - Ocala, Florida
  - Orlando, Florida
  - South Miami, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Gurnee, Illinois
  - Wichita, Kansas
  - Lexington, Kentucky
  - Boston, Massachusetts
  - South Dartmouth, Massachusetts
  - Brooklyn Center, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Edison, New Jersey
  - Endwell, New York
  - Burlington, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Yukon, Oklahoma
  - Bensalem, Pennsylvania
  - Mt. Pleasant, South Carolina
  - Nashville, Tennessee
  - Fort Worth, Texas
  - New Braunfels, Texas
  - San Antonio, Texas
  - West Jordan, Utah
  - Wauwatosa, Wisconsin